CLINICAL TRIAL: NCT04409535
Title: Effects of the COVID-19 Health Emergency on the Biopsychosocial Health of Rural Residents of New Mexico Using Mixed Methods Research
Brief Title: Effects of the COVID-19 Health Emergency on Biopsychosocial Health
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Carla S. Wilhite, Assistant Professor, University of New Mexico
Other Study IDs: 20-266
Record Dates: First submitted 2020-05-11; First posted 2020-06-01 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Activities; Mental Health Issue; Life Style
Keywords: Quality of Life; Rural Community; COVID-19
MeSH Terms: conditions — Motor Activity; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rural Living Community Member: Adult residents of a New Mexico rural county (as federally designated)
  Interventions: Other: WHOQOL-BREF survey
- Urban/Suburban Living Community Member: Comparison group: adult resident of a New Mexico urban/suburban city or town (as federally designated)
  Interventions: Other: WHOQOL-BREF survey

INTERVENTIONS:
Other: WHOQOL-BREF survey — Participants will be surveyed and interviewed about their perceptions regarding COVID-19 health emergency
  Other Names: Personal Interview

SUMMARY:
There is a critical need to determine the impact of the COVID-19 emergency on the comprehensive well-being of people as they are living through the emergency and sequelae of the emergency period. The research team is requesting National Institutes of Health funding with the goal to investigate rural vs. urban living people's response to the crisis and its impact using mixed methods research.

DETAILED DESCRIPTION:
The state of New Mexico and the entire nation have entered an unprecedented health emergency created by the COVID-19 virus; affecting the lives of all people, many of whom were significantly unprepared for the disruptions the emergency created in daily life. Rural residents are at increased risk from effects of the emergency due to numerous disadvantages as compared to urban living people (i.e. critical care access, food insecurity, social isolation). Very little is known about how people are living through a national emergency event affecting all people of the nation. Therefore, a significant gap in knowledge exists: 1. How are rural-living vs. urban-living people responding physically and mentally to the crisis? 2. What strategies of resilience are employed by people living in rural vs. urban counties? 3. What are perceptions of access to critical supplies and services in urban vs. rural counties; 4. How is the availability and use of technology used for news, reliable information, and communication? and 5. Use of time: what alterations in daily life self-care, care of others, commerce, and valued routines in urban vs. rural counties are occurring?

ELIGIBILITY:
Inclusion Criteria:

* Urban and rural living residents of New Mexico, any gender, gender identity, any ethnic origin, any health status (healthy, chronic, disabled), and adult age from 18-85

Exclusion Criteria:

* Non-New Mexico residents, adults unable to give consent due to cognition or incarceration status

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urban or rural living residents of New Mexico currently living under the "stay at home" emergency secondary to COVID-19
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
World Health Organization Quality of Life-Brief Scale | From enrollment until post-event (Feb. 2021)
  participant responses about quality of life during COVID-19 emergency

SECONDARY OUTCOMES:
Open-ended Interview | From enrollment until post-event (Feb. 2021)
  Participants responses to open-ended interview questions regarding alteration in daily life routines

CONTACTS AND LOCATIONS:
Overall Officials: Carla Wilhite, DOT, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Department of Pediatrics, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, aggregated data will be available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: March 2021 (tentative) and will be available for three years
Access Criteria: Written request from other academic research university

DOCUMENTS (3):
  • Study Protocol (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT04409535/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT04409535/SAP_001.pdf
  • Informed Consent Form (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT04409535/ICF_002.pdf